CLINICAL TRIAL: NCT03628573
Title: Investigating Biomarkers in Inpatients With Depression Receiving Accelerated Repetitive Transcranial Magnetic Stimulation (rTMS)
Brief Title: Biomarkers in Depressed Inpatients Receiving Accelerated rTMS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Fidel Vila-Rodriguez, Dr. Fidel Vila-Rodriguez, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H14-03368
Record Dates: First submitted 2015-12-02; First posted 2018-08-14 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Depression
Keywords: rTMS; Depression; Theta Burst Stimulation; Inpatients; Biomarkers
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intermittent Theta burst stimulation. (Other): Procedure: repetitive transcranial magnetic stimulation (iTBS) to the left Dorsolateral Prefrontal Cortex; 3 sessions per day, for 20 days.
  Interventions: Device: repetitive transcranial magnetic stimulation (MagPro X100).; Device: Intermittent Theta burst stimulation ( iTBS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (MagPro X100). — accelerated rTMS.
Device: Intermittent Theta burst stimulation ( iTBS)

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is an emerging treatment for medically refractory major depressive disorder (MDD), and involves direct stimulation of cortical neurons using externally applied, powerful, focused magnetic field pulses. rTMS consistently achieves response rates of 50-55% and remission rates of 30-35% in medically refractory MDD patients. However, the vast majority of studies have focused its use in outpatient samples. This study will address whether accelerated rTMS (intermittent Theta Burst Stimulation (iTBS)) can speed up the response rate and shorten length of stay in hospital for inpatients, and which biological traits may predict response.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a highly prevalent and disabling disorder with substantial societal cost; furthermore, the costs associated to MDD increase substantially when it requires hospital admission. Among Neurological, Mental and Substance Use (NMS) disorders, depression is the number one cause of disability worldwide. Considering this high increase in prevalence, in addition to the limited efficacy of current treatments, with only 30-40% of patients achieving remission after an initial treatment, the illness burden attributable to NMS is projected to increase during the next decade. In Ontario alone, $12.5 billion a year is attributed to mood disorder related costs. Unfortunately, research into the treatment and prevention of mental illness is disproportionately low relative to the disease burden. Approved by Health Canada for MDD in 2002, repetitive transcranial magnetic stimulation (rTMS) is an emerging treatment for medically refractory major depressive disorder (MDD). rTMS involves direct stimulation of cortical neurons using externally applied, powerful, focused magnetic field pulses. Dozens of studies and several meta-analyses over the last 15 years have shown that rTMS of the dorsolateral prefrontal cortex (DLPFC) produces statistically significant improvements in MDD, even when medications have failed. In the most recent generation of randomized controlled trials, rTMS consistently achieves response rates of 50-55% and remission rates of 30-35% in medically refractory MDD patients. However, the vast majority of studies have focused on its used in outpatient samples. Furthermore, the few studies that have investigated its used in inpatient samples have demonstrated similar efficacy rates than medications using the conventional 10 Hz rTMS protocol. No study, has addressed the question whether rTMS can speed up the response rate, and shorten length of stay in hospital, nor what are the biomarkers of treatment response to rTMS in inpatient population. Conventional rTMS protocols, as used in the major trials in the USA that secured FDA approval in 2008, applied 3000 pulses of unpatterned, 10 Hz stimulation administered over 37.5 minutes. These protocols limit the number of patients who can be treated with a single machine to approximately 10 per day, thus perpetuating the high cost of treatment. In contrast, iTBS has been shown to have induce neuroplasticity, effective in MDD, and only requires 3 minutes to administer, making it a feasible option for multiple treatments per day, particularly in inpatient populations.

Therefore, addressing the question of biomarkers in inpatient population suffering MDD and whether improvement can be accomplished in only 3 weeks is a critical question with very direct impact and translation to clinical care.

HYPOTHESES:

1. Response to an index course of accelerated Left-iTBS 3 treatments per day will be associated with associated with increased activation of frontal regions in functional Near Infrared Spectroscopy (fNIRS) and electroencephalogram (EEG) (increase cerebral blood flow to left DLPFC, and decrease in alpha power in left DLPFC), and decrease of inflammatory biomarkers.
2. Depression scores on Hamilton Depression Ration Scale (HDRS)-17 will decrease by at the end of second week of treatment, in 50% of the sample.

OBJECTIVES:

1. To investigate neurophysiological and inflammatory biomarkers in inpatients with depression treated with accelerated rTMS.
2. To investigate the speed in reduction of symptoms to accelerated rTMS in MDD in inpatient setting.

PROCEDURES:

The entire study will recruit a total of 50 inpatients. Patients meeting symptomatic criteria for a depressive episode will receive Left-iTBS 3 treatments per day, 45 to 1 hour apart, for a total of 20 consecutive days. Patients will undergo motor threshold testing to determine the appropriate site and strength of stimulation according to standard methods then begin treatment. Measure will also include electroencephalography (EEG), near infrared spectroscopy (fNIRS), a blood draw, and cognitive testing, questionnaires. The treatment phase will last 20 days. Treatment will be administered daily in the morning (60 treatments total).

ELIGIBILITY:
Inclusion Criteria:

1. are inpatients at the time of enrolment;
2. are capable to consent to treatment;
3. are experiencing a major depressive episode that is deemed as the principal concern during the current admission; (3.1) Those who are experiencing a bipolar depressive episode, are on a mood stabilizer;
4. are between the ages of 19 and 65 years;
5. have a score >= 18 on the HDRS-17 item within 2-days prior to initiating TBS;
6. have had no increase or initiation of antidepressant medication in the 4 weeks prior to initiation of TMS (according to clinical judgment);
7. able to adhere to the treatment schedule;
8. pass the TMS adult safety screening (TASS) questionnaire.

Exclusion Criteria:

1. have a history of substance dependence or abuse within the last 3 months;
2. have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump;
3. have active suicidal intent;
4. are experiencing psychosis;
5. are pregnant;
6. have failed a course of electroconvulsive therapy in the current depressive episode or previous episode;
7. have received rTMS for any previous indication due to the potential compromise of expectancy effects;
8. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, history of epilepsy, cerebral aneurysm, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than 5 minutes;
9. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
10. have a clinically significant laboratory abnormality, in the opinion of the one of the principal investigators;
11. are currently (or in the last 4 weeks) taking lorazepam greater than 4 mg daily (or equivalent) or currently taking any dose of an anticonvulsant (those with unipolar depression).

    Note: those with Bipolar depression are allowed to be on mood stabilizers.
12. have a non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
To measure changes in EEG power, before and after 3 weeks of treatment with Theta Burst Stimulation in inpatients with depression. | At baseline, 14 days, 2 weeks post-treatment
To measure changes in cerebral blood flow before and after 3 weeks of treatment with Theta Burst Stimulation in inpatients with depression. | At baseline, 14 days, 2 weeks post-treatment
To measure changes in inflammatory markers before and after 3 weeks of treatment with Theta Burst Stimulation in inpatients with depression. | At baseline, 2 weeks post-treatment

SECONDARY OUTCOMES:
Change in depression score measured by MADRS over the course of Theta Burst Stimulation to accelerated rTMS in MDD in inpatient setting. | At baseline, 5 days, 12 days, 20 days, 2 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fidel Vila-Rodriguez, MD, Principal Investigator — University of British Columbia